CLINICAL TRIAL: NCT04344951
Title: Chloroquine Phosphate Against Infection by the Novel Coronavirus SARS-CoV-2 (COVID-19): The HOPE Open-Label, Non Randomized Clinical Trial
Acronym: HOPE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No clinical efficacy against SARS-CoV-2 recorded
Sponsor: Uni-Pharma Kleon Tsetis Pharmaceutical Laboratories S.A. (Industry)
Collaborators: Athens General Hospital Hippokrateio (Unknown); Sotiria Thoracic Diseases Hospital of Athens (Other); Sismanoglio General Hospital (Other); Divine Providence Hospital Pammakaristos (Unknown); AHEPA University Hospital (Other); University Hospital, Ioannina (Other); Corfu General Hospital Agia Irini (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UNIKINON-01/HOPE
Record Dates: First submitted 2020-04-06; First posted 2020-04-14 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Pneumonia, Viral; Covid-19
Keywords: COVID-19; Pneumonia; Chloroquine phosphate; SARS-CoV-2
MeSH Terms: conditions — Pneumonia, Viral; COVID-19; Pneumonia | interventions — chloroquine diphosphate

STUDY DESIGN:
Intervention Model Description: Prospective, open label, Phase II study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UNIKINON (Chloroquine phosphate) (Experimental): Once a patient is considered eligible for the study, they will receive oral chloroquine phosphate. The total duration of treatment will be 7 days. The dosage will be 500mg every 12 hours. It is clarified that any other treatment at the discretion of the therapist is permitted except for the administration of hydroxychloroquine.
  Interventions: Drug: UNIKINON (Chloroquine phosphate) 200mg tablets

INTERVENTIONS:
Drug: UNIKINON (Chloroquine phosphate) 200mg tablets — Two and a half tablets (500mg) twice daily for seven days.

SUMMARY:
This is an open label clinical study to evaluate the activity of chloroquine phosphate in patients with SARS-CoV-2 virus infection. The study aims to document possible prevention of pneumonia in patients staying at home and in improving the symptoms of SARS-CoV-2 pneumonia in patients who will be hospitalised.

DETAILED DESCRIPTION:
Humanity has been experiencing a new pandemic of the SARS Coronavirus-19 virus (SARS-CoV-2) since December 2019, causing the disease known as COVID-19. As of March 23, 2020, there have been 382,341 documented episodes of infection worldwide, of which 16,567 have died. An important limitation in the treatment of the disease is the absence of drugs with known antiviral activity against SARS-CoV-2. Recent data suggest that chloroquine has sufficient in vitro activity against the SARS-CoV-2 virus by inhibiting virus entry into cells. It has recently been described that hydroxychloroquine significantly reduces the percentage of patients who have positive sputum in the SARS-CoV-2 virus within 6 days. However, the clinical efficacy of the drug has not been described and it has significant side effects, including more than 10% anorexia, headache, blurred vision, diarrhea or vomiting, and myocardiotoxicity. The frequency of adverse effects of chloroquine in combination with the well-known in vitro activity of chloroquine have led to the design of clinical trials around the world to document the benefits of its use. The present study will evaluate the activity of chloroquine phosphate in patients with SARS-CoV-2 virus infection.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Both genders
* For women of childbearing age, they should use or be willing to use a double contraceptive method during the study. A urine pregnancy test to exclude pregnancy will be performed prior to study initiation.
* Written consent after information provided by the patient or the legal representative in the event that the patient cannot consent.
* Upper respiratory or lower respiratory tract infection, as in Annexes II and III respectively.
* Positive respiratory secretion test for SARS-CoV-2 virus by molecular techniques or positive blood IgM titers.

Exclusion Criteria:

* Under 18 years of age
* Denial of written consent
* Any patient case where it has been decided not to rejuvenate
* Serum AST values greater than 5 times the upper normal range
* QTc interval in rest electrocardiogram greater than 500msecs
* Pregnancy or lactation. Urgent pregnancy test to exclude pregnancy before inclusion in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
50% reduction in symptom score for patients with lower respiratory tract infection | Day 8 visit from study initiation
  Achieving 50% reduction in symptom score for patients with lower respiratory tract infection on day 8 visit from study initiation.
Lack of progression for patients with upper respiratory tract infection | Day 8 visit from study initiation
  Lack of progression to lower respiratory tract infection in patients enrolled in the study due to upper respiratory tract infection on day 8 visit from study initiation.

SECONDARY OUTCOMES:
Comparison of the primary endpoint with respective patients not receiving the treatment | Day 14 visit from study initiation
  Lower respiratory tract infection rating takes place. The symptoms checked are: Cough, Chest pain, Dyspnea, expectoration. For each symptom score is given from 0 to 3 depending on the intensity and they are summed.
Serious respiratory failure until day 14. This will be compared with respective patients not receiving the treatment. | Day 14 visit from study initiation
  It is defined as the presence of both of the following:
  * Respiratory quotient (pO2 / FiO2) less than 150
  * Need for treatment with CPAP or mechanical ventilation
Frequency of AEs and SAEs | Day 14 visit from study initiation
  Frequency of AEs and SAEs

CONTACTS AND LOCATIONS:
Overall Officials: Helen Sambatakou, MD, Principal Investigator — Athens General Hospital "Hippokrateio", 2nd department of Pathology; Nikolaos Koulouris, MD, Principal Investigator — Athens General Hospital of Thoracic Diseases "SOTIRIA", 1st University Pulmonary Clinic; Garyfallia Poulakou, MD, Principal Investigator — Athens General Hospital of Thoracic Diseases "SOTIRIA", 3rd University Pathology Clinic; Malvina Lada, MD, Principal Investigator — General Hospital of Athens "Sismanoglio", 2nd Department of Pathology; Ioannis Baraboutis, MD, Principal Investigator — Divine Providence Hospital "Pammakaristos", Pathology Department; Symeon Metallidis, MD, Principal Investigator — University General Hospital of Thessaloniki AHEPA, 1st University Pathology Clinic; Haralambos Milionis, MD, Principal Investigator — University General Hospital of Ioannina, 1st University Pathology Clinic; Ilias Papanikolaou, MD, Principal Investigator — Corfu General Hospital Agia Irini, Pulmonary Clinic
Locations (8):
- Greece (8):
  - Divine Providence Hospital "Pammakaristos", Athens
  - Athens General Hospital "Hippokrateio", Athens
  - Athens General Hospital of Thoracic Diseases "SOTIRIA", 1st University Pulmonary Clinic, Athens
  - Athens General Hospital of Thoracic Diseases "SOTIRIA", 3rd University Pathology Clinic, Athens
  - Corfu General Hospital Agia Irini, Corfu
  - University General Hospital of Ioannina, Ioannina
  - General Hospital of Athens "Sismanoglio", Marousi
  - University General Hospital of Thessaloniki AHEPA, Thessaloniki

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Arabi YM, Murthy S, Webb S. COVID-19: a novel coronavirus and a novel challenge for critical care. Intensive Care Med. 2020 May;46(5):833-836. doi: 10.1007/s00134-020-05955-1. Epub 2020 Mar 3. No abstract available. PMID 32125458
- [Result] Devaux CA, Rolain JM, Colson P, Raoult D. New insights on the antiviral effects of chloroquine against coronavirus: what to expect for COVID-19? Int J Antimicrob Agents. 2020 May;55(5):105938. doi: 10.1016/j.ijantimicag.2020.105938. Epub 2020 Mar 12. PMID 32171740
- [Result] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204